CLINICAL TRIAL: NCT05562232
Title: The Effect of Creatine Monohydrate on Persistent Post-concussive Symptoms - a Pilot Study Protocol
Brief Title: The Effect of Creatine Monohydrate on Persistent Post-concussive Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Michael Haurum Marcussen, Dr., Psychiatric Research Unit, Region Zealand, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRURegionZealand4
Record Dates: First submitted 2022-09-14; First posted 2022-09-30 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Mild Traumatic Brain Injury; Concussion, Brain
Keywords: Concussion; Mild traumatic brain injury; Creatine monohydrate; Persistent post-concussive symptoms
MeSH Terms: conditions — Brain Concussion | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention group (Experimental): Creatine monohydrate administered once a day for seven weeks - with 5 g/day for the entire period.
  Interventions: Dietary Supplement: Creatine Monohydrate
- Control group (No Intervention): The control group will receive standard care. However, to our knowledge there is no common accepted description of a standard care in the literature. In general, these participants will be advised to keep themselves as asymptomatic as possible throughout the entire seven weeks, and besides that live as normal a life as they can.
- Placebo (Placebo Comparator): Powdered Sugar administered once a day for seven weeks - with 5g/day for the entire period.
  Interventions: Dietary Supplement: Creatine Monohydrate

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — Follows
  Arms: Intervention group; Placebo

SUMMARY:
The purpose of this study, is to investigate whether creatine monohydrate as a supplement reduces the number and severity of symptoms in patients with persistent post-concussive symptoms through self-reported post-concussion symptoms questionnaires.

DETAILED DESCRIPTION:
Mild traumatic brain injury (mTBI), which throughout the literature is used interchangeably with concussion, is a problem of public concern. It is estimated that between 0.6 % and 1.2 % of the general population will suffer an mTBI each year which equals to 48-96 millions of people on a world scale. Out of these, an estimated 10-30 % of the patients, will suffer from persistent PPCS. These symptoms typically includes headache, poor concentration, memory problems, fatigue, sleep difficulties, dizziness, irritability, feeling nervous or anxious. PPCS has proven to be not only a health problem, but also a socioeconomical problem. Data has showed that salary in Denmark five years after a concussion decreased 4.2 %, with an increased risk of losing ones job. At the moment no single treatment option is available with guaranteed success, and therefore nutritional supplements are a possibility.

The nutritional supplement CrM is one of the most popular ergogenic aids on the market among professional and amateur athletes. It is mostly used in the development of muscle mass, as creatine is primarily located skeletal muscle. Roughly five percent of the body's creatine is distributed in the brain and testicles. As mTBI's also see a change in the metabolism of the brain, creatine supplementation might be beneficial for patients with PPCS. This is further supported by a newly conducted study, that creatine supplementation may reduce the severity of mild concussion in animal models.

Furthermore, as the enzyme Creatine Kinease (CK), which is involved in ATP energy system, also has a brain specific isoform (BB-CK), creatine may be a relevant part of the energy system of the central nervous system (CNS). In addition evidence points towards creatine supplementation can increase cellular energy availability. It has been reported to increase brain phosphocreatine content by as much as 15 %, which in turn improves the metabolic processes of the brain.

CrM has been described to be a potent anti-inflammatory molecule. It has been shown to reduce the cytotoxic effects in oxidatively-injured cells without affecting antioxidant enzyme activities, and has been shown to inhibit reactive oxygen species-induced formation of mitochondrial permeability transition pores in the liver mitochondria of mice. At the same time, concussion seems to increase inflammation in the brain, and this inflammation has been hypothesized to correlate with the symptomatology and duration. And even though research in the area of recovery is still scarce, neuroinflammation seems to play a vital role in the pathophysiology of concussions. This warrants hopes of a decrease in post-concussive symptoms.

Other studies have indicated an improvement of cognitive functions, including fatigue, working memory and mood state. All symptoms related to PPCS. Additionally evidence points towards creatine supplementation can help with chronic fatigue, depression and anxiety. All this points towards CrM being helpful in the treatment of PPCS.

Currently there is not viable treatment option for these patients, but if the intervention shows positive results, patients suffering from PPCS would be able to improve on their symptoms, relatively easy and cheap. They would have a go-to supplement, that would make it possible for them to get a normal day, without any of the symptoms connected to PPCS.

The pilot study will be performed as a randomized controlled trial in accordance with the Spirit Guidelines. The study is expected to include a convenience sample of 45 patients. The patients will randomly be allocated to either a control group, placebo group or intervention group, with 15 patients in each. The study will be double blinded, i.e., the participants and personel not knowing which group the patients will be allocated to. Furthermore, the process of randomization will consist of a nutritionist not otherwise associated with the study, randomly allocating each participant in a group, until sample size is reached. The person in charge of this, will also be distributing either the placebo or the CrM to the participants in each of these groups.

CG will not receive any treatment other than usual treatment. PLA and INT will both receive a powder, that has to be ingested. PLA will receive a powder similar in looks to CrM, but with no apparent nutritional value, while INT will receive CrM.

As both PLA and INT are the interventions, they will follow the same protocol for ingestion: 5 grams pr day in seven weeks. All 5 grams will be ingested at once. This protocol has been chosen instead of the more common 0.3 g/day for the first week, ingested over five times during the day. In other studies on CrM and the brain, this have been the chosen strategy also. But studies on CrM in the muscles show, that both protocols illicit the same response with 28 days, and the loading phase is not required. Furthermore, some studies have used this protocol with creatine supplementation, and found increased cognitive function. Our reason for choosing 5 g/day in seven weeks, is to increase the chances of compliance, and decrease the risks of discomfort with to high an intake of CrM. An intake five times a day for the first week, is demanding, and will most likely get some participants to quit the study.

At the mid phase of the study, all baseline measurements will be done again. The length of the intervention is seven weeks. After the seven weeks, all baseline measurements will be done again. And a week after last ingestion, the measurements will be done one last time. At the week eight appointment, every participant will have to answer whether they thought they were getting placebo or CrM. This is done in order to figure out how big an effect placebo have on the results.

The control group will receive standard care. However, to our knowledge there is no common accepted description of a standard care in the literature., In general, these participants will be advised to keep themselves as asymptomatic as possible throughout the entire seven weeks, and besides that live as normal a life as they can.

The study population will be patients with persistent post-concussive symptoms between six and twelve months at start of participation. Participants will be recruited through social media and fourteen neurological outpatient clinics located in Denmark. At the start of the study, participants will have to be between 25 and 35 years of age. This will make the population a homogenous age group, and we will avoid physical and cognitive challenges related to early childhood and adolescents, as well as avoiding the degeneration in physical capacities that begin at approximately the age of 35, as well as the cognitive decline around the same time.

The anthropometrics of the participants will consist of age (years), gender (male/female), height (cm), bodymass (kg), period with PPCS (months), concussion history (yes/no), if yes, then how many (number), and training status (hours/week).

ELIGIBILITY:
Inclusion Criteria:

* Have had PPCS for a minimum of six months and a maximum of 18 months at the start of the study.
* Being between 20 and 45 years of age

Exclusion Criteria:

* Elite athletes, as well as people who in general is physical active, at an intensity of moderat to high, for more than ten hours a week on average.
* Participation in other interventions/treatment that could affect this study
* Have had PPCS in:
* =<6 months
* =>18 months
* Pregnant

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Post-Concussion Symptoms at 7 weeks | Baseline, 3 weeks and 7 weeks (follow-up)
  Rivermead Post-Concussion Symptom Questionnaire

SECONDARY OUTCOMES:
Change from Baseline Body weight at 7 weeks | Baseline, 3 weeks and 7 weeks (follow-up)
  As we are using a dietary supplement as our intervention, following participants body weight in kg throughout the intervention is necessary in order to know if changes in body weight have any effect on our results.

OTHER OUTCOMES:
Height | Baseline
  Descriptive measurement
Training status | Baseline
  To determine if the participants are at the same initial training status.
Period with PPCS | Baseline
  To assess persistent post-concussive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marcussen, Dr., Principal Investigator — University of Southern Denmark (SDU), Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Background] McCrory P, Meeuwisse W, Dvorak J, Aubry M, Bailes J, Broglio S, Cantu RC, Cassidy D, Echemendia RJ, Castellani RJ, Davis GA, Ellenbogen R, Emery C, Engebretsen L, Feddermann-Demont N, Giza CC, Guskiewicz KM, Herring S, Iverson GL, Johnston KM, Kissick J, Kutcher J, Leddy JJ, Maddocks D, Makdissi M, Manley GT, McCrea M, Meehan WP, Nagahiro S, Patricios J, Putukian M, Schneider KJ, Sills A, Tator CH, Turner M, Vos PE. Consensus statement on concussion in sport-the 5th international conference on concussion in sport held in Berlin, October 2016. Br J Sports Med. 2017 Jun;51(11):838-847. doi: 10.1136/bjsports-2017-097699. Epub 2017 Apr 26. No abstract available. PMID 28446457
- [Background] Cassidy JD, Carroll LJ, Peloso PM, Borg J, von Holst H, Holm L, Kraus J, Coronado VG; WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. Incidence, risk factors and prevention of mild traumatic brain injury: results of the WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. J Rehabil Med. 2004 Feb;(43 Suppl):28-60. doi: 10.1080/16501960410023732. PMID 15083870
- [Background] Langer L, Levy C, Bayley M. Increasing Incidence of Concussion: True Epidemic or Better Recognition? J Head Trauma Rehabil. 2020 Jan/Feb;35(1):E60-E66. doi: 10.1097/HTR.0000000000000503. PMID 31246881
- [Background] Makdissi M, Schneider KJ, Feddermann-Demont N, Guskiewicz KM, Hinds S, Leddy JJ, McCrea M, Turner M, Johnston KM. Approach to investigation and treatment of persistent symptoms following sport-related concussion: a systematic review. Br J Sports Med. 2017 Jun;51(12):958-968. doi: 10.1136/bjsports-2016-097470. Epub 2017 May 8. PMID 28483928
- [Background] Levin HS, Diaz-Arrastia RR. Diagnosis, prognosis, and clinical management of mild traumatic brain injury. Lancet Neurol. 2015 May;14(5):506-17. doi: 10.1016/S1474-4422(15)00002-2. Epub 2015 Mar 20. PMID 25801547
- [Background] Fallesen P, Campos B. Effect of concussion on salary and employment: a population-based event time study using a quasi-experimental design. BMJ Open. 2020 Oct 21;10(10):e038161. doi: 10.1136/bmjopen-2020-038161. PMID 33087373
- [Background] Kreider RB, Kalman DS, Antonio J, Ziegenfuss TN, Wildman R, Collins R, Candow DG, Kleiner SM, Almada AL, Lopez HL. International Society of Sports Nutrition position stand: safety and efficacy of creatine supplementation in exercise, sport, and medicine. J Int Soc Sports Nutr. 2017 Jun 13;14:18. doi: 10.1186/s12970-017-0173-z. eCollection 2017. PMID 28615996
- [Background] Romeu-Mejia R, Giza CC, Goldman JT. Concussion Pathophysiology and Injury Biomechanics. Curr Rev Musculoskelet Med. 2019 Jun;12(2):105-116. doi: 10.1007/s12178-019-09536-8. PMID 30820754
- [Background] Kreider RB, Stout JR. Creatine in Health and Disease. Nutrients. 2021 Jan 29;13(2):447. doi: 10.3390/nu13020447. PMID 33572884
- [Background] Smith RN, Agharkar AS, Gonzales EB. A review of creatine supplementation in age-related diseases: more than a supplement for athletes. F1000Res. 2014 Sep 15;3:222. doi: 10.12688/f1000research.5218.1. eCollection 2014. PMID 25664170
- [Background] Lowe MT, Faull RL, Christie DL, Waldvogel HJ. Distribution of the creatine transporter throughout the human brain reveals a spectrum of creatine transporter immunoreactivity. J Comp Neurol. 2015 Apr 1;523(5):699-725. doi: 10.1002/cne.23667. Epub 2014 Sep 12. PMID 25159005
- [Background] Whyte MP, Chines A, Silva DP Jr, Landt Y, Ladenson JH. Creatine kinase brain isoenzyme (BB-CK) presence in serum distinguishes osteopetroses among the sclerosing bone disorders. J Bone Miner Res. 1996 Oct;11(10):1438-43. doi: 10.1002/jbmr.5650111010. PMID 8889843
- [Background] Roschel H, Gualano B, Ostojic SM, Rawson ES. Creatine Supplementation and Brain Health. Nutrients. 2021 Feb 10;13(2):586. doi: 10.3390/nu13020586. PMID 33578876
- [Background] Hanna-El-Daher L, Braissant O. Creatine synthesis and exchanges between brain cells: What can be learned from human creatine deficiencies and various experimental models? Amino Acids. 2016 Aug;48(8):1877-95. doi: 10.1007/s00726-016-2189-0. Epub 2016 Feb 10. PMID 26861125
- [Background] Sestili P, Martinelli C, Bravi G, Piccoli G, Curci R, Battistelli M, Falcieri E, Agostini D, Gioacchini AM, Stocchi V. Creatine supplementation affords cytoprotection in oxidatively injured cultured mammalian cells via direct antioxidant activity. Free Radic Biol Med. 2006 Mar 1;40(5):837-49. doi: 10.1016/j.freeradbiomed.2005.10.035. Epub 2005 Nov 2. PMID 16520236
- [Background] O'Gorman E, Beutner G, Dolder M, Koretsky AP, Brdiczka D, Wallimann T. The role of creatine kinase in inhibition of mitochondrial permeability transition. FEBS Lett. 1997 Sep 8;414(2):253-7. doi: 10.1016/s0014-5793(97)01045-4. PMID 9315696
- [Background] Watanabe A, Kato N, Kato T. Effects of creatine on mental fatigue and cerebral hemoglobin oxygenation. Neurosci Res. 2002 Apr;42(4):279-85. doi: 10.1016/s0168-0102(02)00007-x. PMID 11985880
- [Background] Rae C, Digney AL, McEwan SR, Bates TC. Oral creatine monohydrate supplementation improves brain performance: a double-blind, placebo-controlled, cross-over trial. Proc Biol Sci. 2003 Oct 22;270(1529):2147-50. doi: 10.1098/rspb.2003.2492. PMID 14561278
- [Background] Avgerinos KI, Spyrou N, Bougioukas KI, Kapogiannis D. Effects of creatine supplementation on cognitive function of healthy individuals: A systematic review of randomized controlled trials. Exp Gerontol. 2018 Jul 15;108:166-173. doi: 10.1016/j.exger.2018.04.013. Epub 2018 Apr 25. PMID 29704637
- [Background] Bakian AV, Huber RS, Scholl L, Renshaw PF, Kondo D. Dietary creatine intake and depression risk among U.S. adults. Transl Psychiatry. 2020 Feb 3;10(1):52. doi: 10.1038/s41398-020-0741-x. PMID 32066709
- [Background] Bender A, Klopstock T. Creatine for neuroprotection in neurodegenerative disease: end of story? Amino Acids. 2016 Aug;48(8):1929-40. doi: 10.1007/s00726-015-2165-0. Epub 2016 Jan 9. PMID 26748651
- [Background] Sowell ER, Thompson PM, Holmes CJ, Jernigan TL, Toga AW. In vivo evidence for post-adolescent brain maturation in frontal and striatal regions. Nat Neurosci. 1999 Oct;2(10):859-61. doi: 10.1038/13154. No abstract available. PMID 10491602
- [Background] Johnson SB, Blum RW, Giedd JN. Adolescent maturity and the brain: the promise and pitfalls of neuroscience research in adolescent health policy. J Adolesc Health. 2009 Sep;45(3):216-21. doi: 10.1016/j.jadohealth.2009.05.016. PMID 19699416
- [Background] Westerstahl M, Jansson E, Barnekow-Bergkvist M, Aasa U. Longitudinal changes in physical capacity from adolescence to middle age in men and women. Sci Rep. 2018 Oct 3;8(1):14767. doi: 10.1038/s41598-018-33141-3. PMID 30283061
- [Background] Peters R. Ageing and the brain. Postgrad Med J. 2006 Feb;82(964):84-8. doi: 10.1136/pgmj.2005.036665. PMID 16461469
- [Background] King NS, Crawford S, Wenden FJ, Moss NE, Wade DT. The Rivermead Post Concussion Symptoms Questionnaire: a measure of symptoms commonly experienced after head injury and its reliability. J Neurol. 1995 Sep;242(9):587-92. doi: 10.1007/BF00868811. PMID 8551320
- [Background] Dechent P, Pouwels PJ, Wilken B, Hanefeld F, Frahm J. Increase of total creatine in human brain after oral supplementation of creatine-monohydrate. Am J Physiol. 1999 Sep;277(3):R698-704. doi: 10.1152/ajpregu.1999.277.3.R698. PMID 10484486
- [Background] Lyoo IK, Kong SW, Sung SM, Hirashima F, Parow A, Hennen J, Cohen BM, Renshaw PF. Multinuclear magnetic resonance spectroscopy of high-energy phosphate metabolites in human brain following oral supplementation of creatine-monohydrate. Psychiatry Res. 2003 Jun 30;123(2):87-100. doi: 10.1016/s0925-4927(03)00046-5. PMID 12850248
- [Background] Antonio J, Candow DG, Forbes SC, Gualano B, Jagim AR, Kreider RB, Rawson ES, Smith-Ryan AE, VanDusseldorp TA, Willoughby DS, Ziegenfuss TN. Common questions and misconceptions about creatine supplementation: what does the scientific evidence really show? J Int Soc Sports Nutr. 2021 Feb 8;18(1):13. doi: 10.1186/s12970-021-00412-w. PMID 33557850
- [Background] Ling J, Kritikos M, Tiplady B. Cognitive effects of creatine ethyl ester supplementation. Behav Pharmacol. 2009 Dec;20(8):673-9. doi: 10.1097/FBP.0b013e3283323c2a. PMID 19773644
- [Background] Harmon KG, Clugston JR, Dec K, Hainline B, Herring S, Kane SF, Kontos AP, Leddy JJ, McCrea M, Poddar SK, Putukian M, Wilson JC, Roberts WO. American Medical Society for Sports Medicine position statement on concussion in sport. Br J Sports Med. 2019 Feb;53(4):213-225. doi: 10.1136/bjsports-2018-100338. PMID 30705232
- [Background] Belanger M, Allaman I, Magistretti PJ. Differential effects of pro- and anti-inflammatory cytokines alone or in combinations on the metabolic profile of astrocytes. J Neurochem. 2011 Feb;116(4):564-76. doi: 10.1111/j.1471-4159.2010.07135.x. Epub 2011 Jan 19. PMID 21143598
- [Background] Balalla S, Krageloh C, Medvedev O, Siegert R. Is the Rivermead Post-Concussion Symptoms Questionnaire a Reliable and Valid Measure to Assess Long-Term Symptoms in Traumatic Brain Injury and Orthopedic Injury Patients? A Novel Investigation Using Rasch Analysis. Neurotrauma Rep. 2020 Aug 11;1(1):63-72. doi: 10.1089/neur.2020.0017. eCollection 2020. PMID 34223531
- [Background] Eyres S, Carey A, Gilworth G, Neumann V, Tennant A. Construct validity and reliability of the Rivermead Post-Concussion Symptoms Questionnaire. Clin Rehabil. 2005 Dec;19(8):878-87. doi: 10.1191/0269215505cr905oa. PMID 16323387
- [Derived] Bodker RL, Marcussen M. Pilot study protocol of a randomized controlled trial for the potential effects of creatine monohydrate on persistent post-concussive symptoms. Front Neurol. 2023 Jul 5;14:1209548. doi: 10.3389/fneur.2023.1209548. eCollection 2023. PMID 37475743